CLINICAL TRIAL: NCT03441386
Title: Acute Physical Exercise Intensity on Cognitive Inhibition and Psychological Well-being in Adolescents
Brief Title: Acute Physical Exercise Intensity on Adolescents Cognitive Function
Acronym: APICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Diego Pastor, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: DPS.EC.02.16
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Cognitive Function and Well-Being

STUDY DESIGN:
Intervention Model Description: Three counterbalanced experimental sessions for the same group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Study (Experimental): Cognitive Responses was analyzed after different intensities physical exercise sessions.
  Interventions: Behavioral: Physical Exercise Session

INTERVENTIONS:
Behavioral: Physical Exercise Session

SUMMARY:
Cognitive function and psychological well-being are two variables related to academic performance. Several studies have shown that these variables are sensitive to acute physical exercise, but it is not known which doses of exercise are the most adaptive. To explore this issue, a quasi-experimental study was conducted with 35 adolescents from three physical education classes. Participants performed three sessions of physical education with different doses of exercise: no exercise, light/moderate exercise, and moderate/vigorous exercise, controlling intensities with accelerometers. All subjects completed the Stroop test (to measure cognitive inhibition) and well-being questionnaires of subjective vitality, positive affect and negative affect before and after each session.

DETAILED DESCRIPTION:
Participants The initial sample comprised 35 students from 2nd grade of high school (19 boys and 16 girls), aged between 16 and 18 years (M =16.49, SD = .79). The students belonged to a public school of a large city in Spain.

Ethical approval and informed consent The experiment was approved by the Ethics Committee of the authors' university and approved by the corresponding academic authority of the high school. All participants signed an informed consent by themselves and their parents.

Measures Measure of Interference Index (Stroop Test). The interference index was calculated from the scores obtained by the participants in the Spanish adaptation of the Stroop test 25 using a pencil-and-paper version.

The test consists of three pages of words and drawings printed in colors that combine in different ways. The first set or page, called Word (W), is made up of the words blue, green, and red, written in black ink on a white background. The second page, called Color (C), presents groups of four Xs (XXXX), printed in one of the above-mentioned colors (blue, red or green). The participants are requested to name the color of the four Xs presented. The last page, called Word-Color (WC) is made up of the names of the colors that appear on page 1, but in ink colors that are incongruent with the printed word. Participants are requested to name the color while inhibiting the reading of the word.

All the pages have 100 items, and each test lasts 45 seconds. The number of hits is added. For this study, we calculated the interference index with the formula, Interference Index = WC - ((WxC)/(W+C)). As indicated by Martín et al. (2012), this index represents the difference between the real performance on page 3 and the expected performance as a function of the hits on pages 1 and 2. Higher values indicate better control of interference.

Measure of psychological well-being Subjective vitality. To measure the students' perception of vitality before and after the three sessions, we used the Subjective Vitality Questionnaire 26, adapted to Spanish by Molina-García, Castillo, and Pablos 27. This questionnaire can be considered as a eudaimonic measure of psychological well-being 17. The questionnaire is made up of 7 items that indicate how the person feels at that moment (e.g., "I am full of energy"). The responses are rated on an 8-point Likert-type scale ranging from 0 (not at all) to 7 (very true). Cronbach's alpha in the different experimental situations ranged from .74 to .82.

Affect. The Spanish version 19 of the short form of the Positive and Negative Affect Schedule 28 was used to measure positive and negative feelings before and after the sessions of physical education. This questionnaire is considered a hedonic measure of well-being. The scale is made up of 9 adjectives, which are grouped into two factors in response to the item "Indicate how you feel right now…". Four of the items represent feelings associated with Positive Affect (glad, happy, content, amused), and five of them represent Negative Affect (depressed, worried, frustrated, angry, unhappy). The responses are rated on an 8-point Likert-type scale ranging from 1 (not at all) to 7 (extremely). Cronbach´s alpha ranged between .76 and. 90 for the two factors in the present study.

Procedure Only the participants who handed in an informed consent signed by themselves, their parents, and the school could participate. They were informed of the confidentiality and anonymity of the results obtained. Although all the adolescents of the three classes that participated in the study underwent all the experimental sessions (as a part of their physical education curriculum), the investigators only measured the students who had handed in the signed informed consent. The final sample (N = 35) was made up of those who participated in all the pre and post-experimental sessions. The investigators counterbalanced the three experimental sessions in the three classes. The participants carried out four sessions (one pre-experimental session and three experimental sessions).

Pre-experimental session. In the first session, the participants completed the socio-demographic data and then carried out a Stroop test training session, before receiving a theoretical physical education class, in order to prevent a possible "learning effect" in test performance. The participants performed a minimum of 2 attempts of each page. When the participants made two attempts with a variability of intra-page hits below 5% with regard to the previous attempt, the training session ended. Thus, the researchers respected individual variability in learning the test. Prior studies have also used this percentage of intra-variability as an indication of stable performance in cognitive inhibition tests 24. Nevertheless, recent studies have shown that the intra-class correlation coefficient of the test in the paper-and-pencil version in Spanish is high when comparing different temporal measures in the same population.

Experimental sessions. The other three sessions consisted of: (a) a 20-min theoretical physical education session, without a physical component, in which the students answered questions about theoretical concepts of training; (b) a session of physical activity of light and moderate intensity, structured as follows: a 5-min warm-up, 20 min of predominantly light and moderate physical activity, and a 5-min cool-off; and (c) a session of physical activity of predominantly moderate and vigorous intensity, with the same structure as before. There was a one-week interval between the sessions. The physical activity sessions were based on aerobics class directed by an instructor.

The duration of the main part of the sessions was established from previous recommendations, which indicate that, for acute sessions of physical activity, the greatest cognitive benefits are obtained with durations of about 20 minutes.

Before and after each session, the adolescents completed the instruments that measured psychological well-being and cognitive interference. The data were collected 15 minutes after the end of each session.

Control of the intensity of the exercise. To control the intensity of the sessions, in addition to measures with accelerometry in each session, the investigators performed a pilot study with 5 adolescents in which they adjusted the intensity of the exercises and the recovery times to ensure that they fulfilled the goals of the session. For this purpose, the investigators used simple aerobic exercises that do not pose any coordination difficulties, and the students followed a monitor's instructions. After adapting the sessions, they were performed in the experimental situation.

The investigators calculated the intensity of the sessions with accelerometry. The investigators used tri-axial GT3X accelerometers that each of the participants wore while performing sessions "b" and "c". The students were shown how to put on and use the accelerometer before beginning the sessions 30. The frequency of time storage was a 1-second "epoch". The investigators ignored periods of use fewer than 15 epochs, and periods of no activity of longer than 1 minute were eliminated from the analysis. The software used for data treatment was ActiLife 6 (Actigraph, Actilife version 6.11.5) and to define the type of activity (light/moderate and moderate/vigorous), the investigators used the cutpoints defined by 31. The investigators chose this author because he clearly and concisely defines the cutpoints as a function of concrete ages. The specific criteria for each age are found in the SAS code available at http://epi.grants.cancer.gov/nhanes_pam/ (National Cancer Institute).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents participants in official Physical Education studies

Exclusion Criteria:

* They must be authorized by their parents.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Cognitive Inhibition Interference Index | 5 minutes after exercise session
  A pen and papel Stroop Test meassure
Subjective Vitality | 5 minutes after exercise session
  Perception of Vitality by Subjective Vitality Questionaire, The questionnaire is made up of 7 items that indicate how the person feels at that moment (e.g., "I am full of energy"). The responses are rated on an 8-point Likert-type scale ranging from 0 (not at all) to 7 (very true).
Affect | 5 minutes after exercise session
  Positive and Negative Affect Schedule, Four of the items represent feelings associated with Positive Affect (glad, happy, content, amused), and five of them represent Negative Affect (depressed, worried, frustrated, angry, unhappy). The responses are rated on an 8-point Likert-type scale ranging from 1 (not at all) to 7 (extremely).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided